CLINICAL TRIAL: NCT02180464
Title: A Phase IIa, 28-day Treatment, Multi-center, Randomized, Comparator-controlled, Observer-blind Trial With Intra-individual Left/Right Comparison to Investigate the Anti-psoriatic Efficacy and the Safety of an LAS41004 Formulation in Comparison to an Active Reference in Patients With Mild to Moderate Plaque Psoriasis
Brief Title: A Intra-individual Comparison to Investigate the Efficacy and the Safety of LAS41004 Formulation in Mild to Moderate Psoriasis
Acronym: Left/Right
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: H 553 000- 1309; 2013-003757-22 (EudraCT Number)
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Psoriasis
Keywords: psoriasis, topical
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LAS41004 (Experimental): Topical application of approximately 2 - 6 mg/cm2 to an area of 20 - 300 cm2, each once daily
  Interventions: Drug: LAS41004; Drug: control
- control (Active Comparator): Topical application of approximately 2 - 6 mg/cm2 of IMPs 1 and 2 to an area of 20 - 300 cm2, each once daily
  Interventions: Drug: LAS41004; Drug: control

INTERVENTIONS:
Drug: LAS41004
Drug: control

SUMMARY:
Proof-of concept study to competitively investigate antipsoriatic efficacy and safety of a LAS41004 formulation vs active control No formal study hypothesis, but descriptive evaluation (PoC).

ELIGIBILITY:
Inclusion Criteria (main):

* mild to moderate stable chronic plaque-type psoriasis with at least two symmetrical lesions with a treatment area of 20 - 300 cm² and a TSS of ≥ 6;

  * female volunteers of childbearing potential* must agree to use appropriate and reliable methods of contraception
  * written informed consent obtained.

Exclusion Criteria (main):

* severe forms of psoriasis or forms of psoriasis other than chronic plaque psoriasis,
* treatment with any locally acting medications which might counter or influence the trial aim within 2 weeks preceding the treatment phase of the trial and during the trial;
* treatment with any systemic medications which might counter or influence the trial aim or phototherapy/PUVA within 4 weeks preceding the treatment phase of the trial and during the trial;
* treatment with vitamin A supplements;
* treatment with any biologics within 3 months preceding the treatment phase of the trial and during the trial, or in the case of ustekinumab, within 6 months;
* treatment with any immunosuppressive medication within 6 months preceding the treatment phase of the trial and during the trial;
* known allergic reactions, irritations or hypersensitivity to the active ingredients
* contraindications according to summary of product characteristics (SmPC) of the active comparator: - pregnancy or nursing;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Total symptom score | day 28 vs baseline
  The primary variable is the TSS. The TSS is calculated by summarizing the individual scores for erythema, scaling and infiltration

SECONDARY OUTCOMES:
Total symtom score (during study performance) | Days 4, 8, 15, and 22
  Change from baseline in the TSS of each treated plaque on Days 4, 8, 15, and 22
Physician's global assessment (PGA) | Days 1, 4, 8, 15, 22 and 29
Physician's global tolerability assessment (PGTA) | 4, 8, 15, 22 and 29

CONTACTS AND LOCATIONS:
Overall Officials: Walter Wigger-Alberti, Dr med, Principal Investigator — bioskin, Hamburg
Locations (1):
- Site 1, Hamburg, Germany